CLINICAL TRIAL: NCT00979225
Title: Improving Quality Through Decision Support for Evidence-Based Pharmacotherapy
Brief Title: Clinical Decision Support for Medication Management and Adherence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency); Northern Piedmont Carolina Community Care Partners (Unknown); North Carolina Division of Medical Assistance (Unknown); North Carolina Office of Rural Health and Community Care (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: Pro00002524; R18HS017072 (AHRQ)
Record Dates: First submitted 2009-09-15; First posted 2009-09-17 (Estimated); Last update posted 2012-12-11 (Estimated); Status verified 2012-12

CONDITIONS: Hypertension; Diabetes Mellitus; Stroke; Myocardial Ischemia; Heart Failure; Asthma
Keywords: health information technology; clinical decision support; medication management; medication adherence
MeSH Terms: conditions — Hypertension; Diabetes Mellitus; Stroke; Myocardial Ischemia; Heart Failure; Asthma; Medication Adherence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Medication report (Experimental): Medication reports delivered to providers at the point of care
  Interventions: Other: Medication Management report
- Med. report plus care manager notices (Experimental): Medication reports delivered to providers at the point of care and notices sent electronically to care managers
  Interventions: Other: Medication Management report; Other: Care manager email notices
- Control (No Intervention)

INTERVENTIONS:
Other: Medication Management report — Patients receive medication management reports delivered to their clinic-based caregivers for pharmacotherapy clinical decision support at point-of-care.
  Other Names: Medication management reports
  Arms: Med. report plus care manager notices; Medication report
Other: Care manager email notices — Community-based care managers receive email notices if the patient has not seen his/her primary care provider in the past 6 months, has low adherence to medications, and has no scheduled appointment.
  Other Names: Care manager notices
  Arms: Med. report plus care manager notices

SUMMARY:
This three-year, grant funded project will be conducted by the Division of Clinical Informatics in the Department of Community and Family Medicine at Duke University Medical Center. The project seeks to improve care quality and safety in an ambulatory care setting through clinical decision support for evidence-based (EB) pharmacotherapy delivered as point-of-care reports to clinic-based practitioners and as population health-based alerts to care managers.

This project will build upon a regional Health Information Exchange (HIE) network created to connect providers serving 37,000 Medicaid beneficiaries from both rural and urban settings in a 5 county region in the Northern Piedmont of North Carolina. This network includes 16 private practices, 3 federally qualified health centers, 5 rural health centers, 3 urgent care facilities, 10 government agencies, 5 hospitals, and 2 cross-disciplinary care management teams.

The proposed information system will be based on an emerging standard for decision support and will utilize routinely available claims and scheduling data in order to serve as a replicable model for broader use of decision support for medication management. Increased availability and use of decision support tools for medication management can be expected to reduce medication errors, improve health care quality at an acceptable cost, and augment disease management for patients and populations.

DETAILED DESCRIPTION:
The study will be conducted in accordance with the following four specific aims:

Aim 1: Expand the functionality of an existing decision support system in use within a regional HIE network to incorporate EB pharmacotherapy guidelines and to promote medication adherence. Primary care clinicians will receive EB pharmacotherapy suggestions and a patient-specific summary of prescription claims data delivered to the point-of-care via fax. Care managers will receive alerts delivered via email to encourage patients to arrange follow-up clinic appointments because of possible medication non-adherence.

Aim 2: Implement and evaluate the impact of the two interventions on adherence to EB pharmacotherapy recommendations among Medicaid patients with high priority conditions as designated by the Institute of Medicine (IOM) in ambulatory care settings through a three-arm randomized controlled trial.

Aim 3: Compare resource utilization and assess the economic attractiveness (cost-savings or cost-effectiveness) of the interventions to promote medication adherence and EB pharmacotherapy.

Aim 4: Disseminate information regarding the development and impact of the interventions through Web teleconferences, professional meetings, educational lectures, and peer review journals.

ELIGIBILITY:
Inclusion Criteria:

* Carolina Access Medicaid patients continuously enrolled for 10 of 12 months prior to August 2009
* Patients assigned to one of 14 participating primary care clinics within the Northern Piedmont Community Care Network
* At least one of six IOM priority conditions: hypertension, diabetes mellitus, stroke, ischemic heart disease, heart failure, or persistent asthma

Exclusion Criteria:

* Patient opted-out

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 5000 (Actual)
Dates: Start 2009-09; Primary Completion 2011-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Rates of aggregate adherence by study group to all applicable pharmacotherapy rules during the study period. | Baseline, 12 months

SECONDARY OUTCOMES:
Rates of adherence to pharmacotherapy rules for a specific therapeutic drug class | Baseline, 12 months
Rates of adherence to pharmacotherapy rules for a specific IOM priority condition. | Baseline, 12 months
Rates of adherence to applicable pharmacotherapy rules 6 months after an intervention was first initiated or could have been initiated for the control arm. | Baseline, 6 months
Rates of adherence by drug class to applicable pharmacotherapy rules 6 months after an intervention was first initiated or could have been initiated for the control arm. | Baseline, 6 months
Rates of adherence by IOM condition to applicable pharmacotherapy rules 6 months after an intervention was first initiated or could have been initiated for the control arm. | Baseline, 6 months
The proportion of email notices that were followed up by a documented care management encounter within 30 days. | 12 months
The proportion of email notices that were followed up by a completed clinic encounter within 60 days. | 12 months
Resource use and medical costs associated with the interventions and their delivery, as well as direct healthcare costs (inpatient and outpatient). | 12 months
Provider satisfaction measured using standard usability survey instruments. | 12 months
Outpatient encounter rates. | Baseline, 12 months
Emergency department encounter rates. | Baseline, 12 months
Inpatient hospitalization rates. | Baseline, 12 months

CONTACTS AND LOCATIONS:
Overall Officials: David F Lobach, MD, PhD, MS, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States